CLINICAL TRIAL: NCT05443113
Title: Early Onset Pectus Excavatum is More Likely to be Part of a Genetic Defect
Brief Title: Young Pectus Excavatum Patients and Genetic Defects
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Ryan Billar, Principal investigator, Erasmus Medical Center
Other Study IDs: MEC-2012-387
Record Dates: First submitted 2022-06-28; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-07

CONDITIONS: Genetic Disease; Pectus Excavatum; Children, Adult
Keywords: Pectus excavatum; Children; Gene; Syndrome
MeSH Terms: conditions — Genetic Diseases, Inborn; Funnel Chest; Syndrome | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children (<11 years) with pectus excavatum: All pediatric PE patients aged younger than 11 years upon first visit of our outpatient clinic
  Interventions: Diagnostic Test: Genetic analysis

INTERVENTIONS:
Diagnostic Test: Genetic analysis — Genetic analysis by geneticists

SUMMARY:
In most pectus excavatum (PE) patients an underlying genetic defect is not found with molecular analysis, as a direct genetic link with PE has yet to be found and because potential underlying genetic disorders are quite rare. Only one-fifth of all PE cases are identified in the first decade of life and thus of congenital origin making younger PE patients a unique patient group. Therefore, the research question is; is early-onset pectus excavatum (PE) more likely to be part of a genetic defect than PE which became apparent during puberty or adolescence?

DETAILED DESCRIPTION:
Importance: In most pectus excavatum (PE) patients an underlying genetic defect is not found with molecular analysis, as a direct genetic link with PE has yet to be found and because potential underlying genetic disorders are quite rare. Only one-fifth of all PE cases are identified in the first decade of life and thus of congenital origin making younger PE patients a unique patient group.

Objective: the investigators hypothesize that early-onset PE is more likely to be part of a genetic defect than PE which became apparent during puberty or adolescence.

Design: Cohort study Setting: Single center Participants: All pediatric PE patients aged younger than 11 years upon first visit of the outpatient clinic of the department of pediatric surgery at the Sophia Children's Hospital - Erasmus Medical Center between 2014 and 2020 were identified and informed consent was obtained for inclusion. Two clinical geneticists performed the anamnesis and physical examination. Molecular analysis was performed based on the differential diagnosis. All young PE patients which have been referred for genetic counseling already, were analyzed retrospectively.

Main Outcome: incidence of genetic defects

ELIGIBILITY:
Inclusion Criteria:

* Patients with pectus excavatum aged younger than 11 years upon first visit of our outpatient clinic

Exclusion Criteria:

* None

Ages: 0 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with pectus excavatum aged younger than 11 years
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Incidence of genetic variations | Baseline
  Incidence of genetic variations in children (<11 years) with pectus excavatum

SECONDARY OUTCOMES:
Evaluation checklist referral of a patient with pectus excavatum for genetic counseling | Through study completion, an average of 1 year
  Evaluation and validation of checklist referral of a patient with pectus excavatum for genetic counseling

CONTACTS AND LOCATIONS:
Overall Officials: René M Wijnen, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
In a scientific journal with a high impact factor
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months

REFERENCES:
- [Derived] Billar R, Heyman S, Kant S, Wijnen R, Sleutels F, Demirdas S, Schnater JM. Early-Onset Pectus Excavatum Is More Likely to Be Part of a Genetic Variation. Eur J Pediatr Surg. 2024 Aug;34(4):325-332. doi: 10.1055/a-2081-1288. Epub 2023 Apr 26. PMID 37100424